CLINICAL TRIAL: NCT05617209
Title: Tissue Factor Pathway Inhibitor (TFPI) and Haemorrhagic Manifestations in Haemophilia A and B Patients
Brief Title: In Vitro Correction of Thrombin Generation by Concizumab (Anti-TFPI) for Severe Hemophilia Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 21CH036
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hemophilia
Keywords: anti-TFPI antibody; thrombin generation; tissue factor concentration
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling: thrombin generation measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe and/or moderate haemophilia A and B: At the end of the consultation and follow-up of the disease, an additional blood sample of 35 ml (8 tubes) will be taken
  Interventions: Other: thrombin generation measurement

INTERVENTIONS:
Other: thrombin generation measurement — Thrombin generation will be measured in Platelets rich plasma induced either by 1 pM TF or 10 pM TF concentration in presence of different aTFPIAb concentrations (0; 0.5 µg/ml; 0.75 µg/ml; 1.0 µg/ml; 2.0 µg/ml; 4.0 µg/ml)

SUMMARY:
Studies have shown, in haemophilia patients, the effectiveness of Anti TFPI antibody (aTFPIAb) to prevent joint and muscular bleeding (tissues poor in Tissue Factor (TF)). However, cases of cerebral thrombosis (tissues rich in TF) have been observed in some patients treated with this antibody. Because an inter-individual variation in thrombin generation correction by aTFPIAb, an aTFPIAb concentration effective at low TF concentration could be at the same time thrombogenic at high TF concentration.

DETAILED DESCRIPTION:
The aim of this study is to determine, for each patient, the minimum concentration of aTFPIAb necessary to restore thrombin generation in the presence of low (1pM) TF concentration and to evaluate at this concentration of aTFPIAb a potential thrombogenic effect in the presence of a high (10pM) TF concentration.

ELIGIBILITY:
Inclusion Criteria:

* Severe or moderate haemophilia A or B patient with FVIII or FIX <5% with or without prophylaxis
* Affiliated or beneficiary of a social security regimen
* Signature of consent

Exclusion Criteria:

* Haemophilia patients aged 12 years or less with a weight less than 30 kg (taking into account the volume of blood collection).
* Patients who received factor VIII concentrates less than 48 hours or factor IX concentrates less than 96 hours prior to the routine blood draw at the Hemophilia Clinic. 96 hours prior to the routine blood draw at the Hemophilia Centre

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Haemophilia A and B patients
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
minimum concentration of anti-TFPI antibody | day 1
  Determine the minimum concentration of anti-TFPI antibody (µg/ml) that normalizes the peak to 1 pM FT

SECONDARY OUTCOMES:
Measurement of the clot structure | day 1
  Measurement of the clot structure (density fibers in g/cm3) by scanning electron microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Tardy, MD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No